CLINICAL TRIAL: NCT04619108
Title: Thrombosomes for Expanded Access Use
Status: No longer available | Type: Expanded Access
Sponsor: Cellphire Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Thrombosomes Expanded Access
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Thrombosomes®

SUMMARY:
Expanded use of Thrombosomes where a clinical trial with Thrombosomes is not an option, Cellphire may elect to provide the Sponsor/Investigator (S/I) expanded access to its investigational product, Thrombosomes.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has presented with WHO Grade 2 or higher bleeding which requires treatment with platelet therapy and there is limited availability of platelets or no other approved clinical alternative.
2. Evidence from the facility blood bank/Medical Director that there are no approved platelet products available for transfusion, or the patient is refractory to platelet transfusion.

   Exclusion Criteria:
3. Clinical circumstances of a history of thrombosis, thromboembolism, or vascular occlusion/ischemia in the prior six months such as defined by a past history of current diagnosis of one or more of the following:

   * arterial or venous thromboembolic disease including acute coronary syndrome
   * peripheral vascular disease
   * arterial or venous thrombosis (except when a prior history of central line thrombosis has resolved)
   * myocardial infarction (MI)
   * stent placement
   * valve replacement and/or repair
   * sinusoidal obstruction syndrome (veno-occlusive disease)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult